CLINICAL TRIAL: NCT01464827
Title: A Randomized, Open-Label, Multicenter Study to Evaluate the Antiviral Activity, Safety, and Pharmacokinetics, of ABT-450 With Ritonavir (ABT-450/r) in Combination With ABT-267 and/or ABT-333 With and Without Ribavirin (RBV) for 8, 12 or 24 Weeks in Treatment-Naïve and Null Responder Subjects With Genotype 1 Chronic Hepatitis C Virus Infection
Brief Title: ABT-450 With Ritonavir and ABT-267 and/or ABT-333 With and Without Ribavirin in Genotype 1 Hepatitis C Virus Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M11-652; 2010-022455-31 (EudraCT Number)
Record Dates: First submitted 2011-09-28; First posted 2011-11-04 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Hepatitis C; Hepatitis C (HCV); Hepatitis C Genotype 1
Keywords: Hepatitis C Genotype 1; Hepatitis C; Interferon-Free; HCV; Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — paritaprevir; dasabuvir; ombitasvir; Ribavirin; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (14):
- Group A (Experimental): Treatment-naïve participants received ABT-450 150 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily for 8 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir
- Group B (Experimental): Treatment-naïve participants received ABT-450 150 mg and ritonavir 100 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily for 12 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: Ribavirin; Drug: Ritonavir
- Group C (Experimental): Treatment-naïve participants received ABT-450 100 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, and ribavirin dosed by weight, twice daily for 12 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir
- Group D (Experimental): Treatment-naïve participants received ABT-450 200 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, and ribavirin dosed by weight, twice daily for 12 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir
- Group E (Experimental): Treatment-naïve participants received ABT-450 150 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, and ABT-333 400 mg twice daily for 12 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ABT-267; Drug: Ritonavir
- Group F (Experimental): Treatment-naïve participants received ABT-450 100 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily for 12 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir
- Group G (Experimental): Treatment-naïve participants received ABT-450 150 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 12 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir
- Group H (Experimental): Treatment-naïve participants received ABT-450 100 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 24 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir
- Group I (Experimental): Treatment-naïve participants received ABT-450 150 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 24 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir
- Group J (Experimental): Participants who were null-responders to previous HCV treatment received ABT-450 200 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, and ribavirin dosed by weight, twice daily, for 12 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir
- Group K (Experimental): Participants who were null-responders to previous HCV treatment received ABT-450 100 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 12 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir
- Group L (Experimental): Participants who were null-responders to previous HCV treatment received ABT-450 150 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 12 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir
- Group M (Experimental): Participants who were null-responders to previous HCV treatment received ABT-450 100 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 24 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir
- Group N (Experimental): Participants who were null-responders to previous HCV treatment received ABT-450 150 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 24 weeks.
  Interventions: Drug: ABT-450; Drug: ABT-333; Drug: ABT-267; Drug: Ribavirin; Drug: Ritonavir

INTERVENTIONS:
Drug: ABT-450 — ABT-450 tablets
Drug: ABT-333 — ABT-333 tablets
  Other Names: Dasabuvir
  Arms: Group A; Group B; Group E; Group F; Group G; Group H; Group I; Group K; Group L; Group M; Group N
Drug: ABT-267 — ABT-267 tablets
  Other Names: Ombitasvir
  Arms: Group A; Group C; Group D; Group E; Group F; Group G; Group H; Group I; Group J; Group K; Group L; Group M; Group N
Drug: Ribavirin — Ribavirin tablets administered at a weight-based dose, between 1,000 to 1,200 mg daily (divided).
  Arms: Group A; Group B; Group C; Group D; Group F; Group G; Group H; Group I; Group J; Group K; Group L; Group M; Group N
Drug: Ritonavir — Ritonavir capsules
  Other Names: Norvir

SUMMARY:
This is a study of combination direct-acting antiviral agents (DAA) with or without ribavirin (RBV) in patients with chronic Hepatitis C Virus (HCV).

DETAILED DESCRIPTION:
A study to evaluate the safety and effectiveness of experimental drugs ABT-450, ABT-267 (also known as ombitasvir), ABT-333 (also known as dasabuvir), ritonavir, and ribavirin in participants with HCV. The study will test the safety and effects of combinations of these drugs in treatments up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-70 years old, inclusive
* Females must be post-menopausal for more than 2 years or surgically sterile or practicing specific forms of birth control
* Chronic hepatitis C virus (HCV), genotype 1 infection
* Treatment-naive OR null-responders to previous treatment with pegylated interferon (pegIFN) and ribavirin (at least 12 weeks of treatment and failure to achieve a 2 log10 HCV RNA decrease at Week 12)
* No evidence of liver cirrhosis

Exclusion Criteria:

* Significant liver disease with any cause other than HCV as the primary cause
* Positive hepatitis B surface antigen and anti-human immunodeficiency virus antibody
* Positive screen for drugs and alcohol
* Significant sensitivity to any drug
* Use of contraindicated or prohibited medications within 1 month of dosing
* Abnormal laboratory tests

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, MD, Study Director — AbbVie
Locations (97):
- United States (60):
  - Site Reference ID/Investigator# 57583, Birmingham, Alabama
  - Site Reference ID/Investigator# 55530, Birmingham, Alabama
  - Site Reference ID/Investigator# 55385, Dothan, Alabama
  - Site Reference ID/Investigator# 55500, Phoenix, Arizona
  - Site Reference ID/Investigator# 55382, Tucson, Arizona
  - Site Reference ID/Investigator# 61042, Bakersfield, California
  - Site Reference ID/Investigator# 43651, Coronado, California
  - Site Reference ID/Investigator# 43652, Costa Mesa, California
  - Site Reference ID/Investigator# 59130, Los Angeles, California
  - Site Reference ID/Investigator# 43565, San Diego, California
  - Site Reference ID/Investigator# 43910, Aurora, Colorado
  - Site Reference ID/Investigator# 43572, Bradenton, Florida
  - Site Reference ID/Investigator# 43584, Ft. Pierce, Florida
  - Site Reference ID/Investigator# 43917, Gainesville, Florida
  - Site Reference ID/Investigator# 55384, Jacksonville, Florida
  - Site Reference ID/Investigator# 44610, Wellington, Florida
  - Site Reference ID/Investigator# 55531, Wellington, Florida
  - Site Reference ID/Investigator# 55536, Zephyrhills, Florida
  - Site Reference ID/Investigator# 55540, Macon, Georgia
  - Site Reference ID/Investigator# 55527, Marietta, Georgia
  - Site Reference ID/Investigator# 44621, Chicago, Illinois
  - Site Reference ID/Investigator# 43576, Indianapolis, Indiana
  - Site Reference ID/Investigator# 55383, Bowling Green, Kentucky
  - Site Reference ID/Investigator# 59124, Shreveport, Louisiana
  - Site Reference ID/Investigator# 43568, Annapolis, Maryland
  - Site Reference ID/Investigator# 55901, Baltimore, Maryland
  - Site Reference ID/Investigator# 43588, Lutherville, Maryland
  - Site Reference ID/Investigator# 55534, Boston, Massachusetts
  - Site Reference ID/Investigator# 43656, Springfield, Massachusetts
  - Site Reference ID/Investigator# 43655, Ann Arbor, Michigan
  - Site Reference ID/Investigator# 43913, Detroit, Michigan
  - Site Reference ID/Investigator# 43587, Saint Paul, Minnesota
  - Site Reference ID/Investigator# 43661, Jackson, Mississippi
  - Site Reference ID/Investigator# 43569, Kansas City, Missouri
  - Site Reference ID/Investigator# 44608, St Louis, Missouri
  - Site Reference ID/Investigator# 55526, Egg Harbor, New Jersey
  - Site Reference ID/Investigator# 43566, Manhasset, New York
  - Site Reference ID/Investigator# 59133, Monticello, New York
  - Site Reference ID/Investigator# 43586, New York, New York
  - Site Reference ID/Investigator# 43573, New York, New York
  - Site Reference ID/Investigator# 55532, Poughkeepsie, New York
  - Site Reference ID/Investigator# 55386, Rochester, New York
  - Site Reference ID/Investigator# 55538, Charlotte, North Carolina
  - Site Reference ID/Investigator# 55522, Fayetteville, North Carolina
  - Site Reference ID/Investigator# 55542, Statesville, North Carolina
  - Site Reference ID/Investigator# 55533, Cincinnati, Ohio
  - Site Reference ID/Investigator# 43665, Cincinnati, Ohio
  - Site Reference ID/Investigator# 43585, Medford, Oregon
  - Site Reference ID/Investigator# 55539, Portland, Oregon
  - Site Reference ID/Investigator# 56622, Philadelphia, Pennsylvania
  - Site Reference ID/Investigator# 43592, Germantown, Tennessee
  - Site Reference ID/Investigator# 55723, Germantown, Tennessee
  - Site Reference ID/Investigator# 43659, Nashville, Tennessee
  - Site Reference ID/Investigator# 59132, Houston, Texas
  - Site Reference ID/Investigator# 43577, San Antonio, Texas
  - Site Reference ID/Investigator# 43662, Annandale, Virginia
  - Site Reference ID/Investigator# 43666, Newport News, Virginia
  - Site Reference ID/Investigator# 43574, Seattle, Washington
  - Site Reference ID/Investigator# 43578, Madison, Wisconsin
  - Site Reference ID/Investigator# 55387, Milwaukee, Wisconsin
- Australia (3):
  - Site Reference ID/Investigator# 44850, Adelaide
  - Site Reference ID/Investigator# 44849, Herston
  - Site Reference ID/Investigator# 44852, Kogarah
- Canada (2):
  - Site Reference ID/Investigator# 44084, Calgary
  - Site Reference ID/Investigator# 43905, Vancouver
- France (8):
  - Site Reference ID/Investigator# 44755, Clichy
  - Site Reference ID/Investigator# 44758, Créteil
  - Site Reference ID/Investigator# 58884, Lyon
  - Site Reference ID/Investigator# 58887, Marseille
  - Site Reference ID/Investigator# 58886, Montpellier
  - Site Reference ID/Investigator# 44754, Paris
  - Site Reference ID/Investigator# 58889, Pessac
  - Site Reference ID/Investigator# 44760, Vandœuvre-lès-Nancy
- Germany (7):
  - Site Reference ID/Investigator# 59304, Berlin
  - Site Reference ID/Investigator# 59303, Berlin
  - Site Reference ID/Investigator# 46103, Frankfurt
  - Site Reference ID/Investigator# 46106, Hamburg
  - Site Reference ID/Investigator# 46102, Hanover
  - Site Reference ID/Investigator# 58922, Kiel
  - Site Reference ID/Investigator# 46105, Würzburg
- Site Reference ID/Investigator# 44847, Auckland, New Zealand
- Puerto Rico (2):
  - Site Reference ID/Investigator# 43672, San Juan
  - Site Reference ID/Investigator# 43675, San Juan
- Spain (8):
  - Site Reference ID/Investigator# 46485, Barcelona
  - Site Reference ID/Investigator# 45363, Barcelona
  - Site Reference ID/Investigator# 45668, Barcelona
  - Site Reference ID/Investigator# 46484, Madrid
  - Site Reference ID/Investigator# 45667, Madrid
  - Site Reference ID/Investigator# 45671, Majadahonda (Madrid)
  - Site Reference ID/Investigator# 46583, Seville
  - Site Reference ID/Investigator# 45405, Valencia
- United Kingdom (6):
  - Site Reference ID/Investigator# 57545, Dundee
  - Site Reference ID/Investigator# 59262, London
  - Site Reference ID/Investigator# 57547, London
  - Site Reference ID/Investigator# 58811, London
  - Site Reference ID/Investigator# 57882, Nottingham
  - Site Reference ID/Investigator# 57543, Southampton

REFERENCES:
- [Derived] Krishnan P, Tripathi R, Schnell G, Reisch T, Beyer J, Irvin M, Xie W, Larsen L, Cohen D, Podsadecki T, Pilot-Matias T, Collins C. Resistance analysis of baseline and treatment-emergent variants in hepatitis C virus genotype 1 in the AVIATOR study with paritaprevir-ritonavir, ombitasvir, and dasabuvir. Antimicrob Agents Chemother. 2015 Sep;59(9):5445-54. doi: 10.1128/AAC.00998-15. Epub 2015 Jun 22. PMID 26100711
- [Derived] Kowdley KV, Lawitz E, Poordad F, Cohen DE, Nelson DR, Zeuzem S, Everson GT, Kwo P, Foster GR, Sulkowski MS, Xie W, Pilot-Matias T, Liossis G, Larsen L, Khatri A, Podsadecki T, Bernstein B. Phase 2b trial of interferon-free therapy for hepatitis C virus genotype 1. N Engl J Med. 2014 Jan 16;370(3):222-32. doi: 10.1056/NEJMoa1306227. PMID 24428468
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 2, open-label, randomized, combination treatment study of multiple doses of ABT-450/ritonavir, and ABT-267 and/or ABT-333 with or without ribavirin in hepatitis C virus (HCV) genotype 1-infected treatment-naïve patients and previous null responders to pegylated interferon (pegIFN) and ribavirin treatment.
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Group G | Group H | Group I | Group J | Group K | Group L | Group M | Group N
Started | 80 | 43 | 39 | 40 | 80 | 39 | 41 | 40 | 40 | 47 | 23 | 23 | 23 | 22
Treated | 80 | 41 | 39 | 40 | 79 | 39 | 40 | 40 | 40 | 45 | 23 | 22 | 23 | 20
Completed | 77 | 36 | 39 | 36 | 72 | 38 | 37 | 37 | 37 | 44 | 21 | 21 | 21 | 19
Not Completed | 3 | 7 | 0 | 4 | 8 | 1 | 4 | 3 | 3 | 3 | 2 | 2 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 2 | 3 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other | 2 | 3 | 0 | 2 | 3 | 0 | 1 | 0 | 3 | 1 | 2 | 0 | 1 | 0
Not completed — Not Treated | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population (participants who received at least 1 dose of direct-acting antiviral agent)
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Group G | Group H | Group I | Group J | Group K | Group L | Group M | Group N | Total
Number analyzed (Participants) | 80 | 41 | 39 | 40 | 79 | 39 | 40 | 40 | 40 | 45 | 23 | 22 | 23 | 20 | 571
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (9.99) | 50.8 (9.84) | 51.1 (8.07) | 49.0 (10.59) | 48.3 (10.53) | 49.4 (9.72) | 51.0 (11.08) | 51.5 (11.95) | 51.5 (9.78) | 50.6 (11.19) | 48.5 (12.91) | 51.2 (12.07) | 51.5 (9.06) | 54.6 (11.78) | 50.3 (10.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 23 | 14 | 20 | 34 | 19 | 16 | 22 | 24 | 18 | 7 | 10 | 8 | 8 | 257
  Male | 46 | 18 | 25 | 20 | 45 | 20 | 24 | 18 | 16 | 27 | 16 | 12 | 15 | 12 | 314

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event was defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this treatment.
  The investigator assessed the relationship of each AE to the use of direct-acting antiviral agents (DAAs) and to ribavirin, and rated the severity of each event as either:
  Mild: The AE was transient and easily tolerated by the participant; Moderate: The AE caused the participant discomfort and interrupted usual activities; Severe: The AE caused considerable interference with the participant's usual activities and could have been incapacitating or life-threatening.
  A serious adverse event was any event that resulted in death, was life-threatening, resulted in or prolonged hospitalization, resulted in a congenital anomaly or persistent or significant disability or was any other important medical event requiring medical or surgical intervention.
Time Frame: From the time of study drug administration until 30 days following discontinuation of study drug administration (up to 28 weeks).
Population: Safety population. Treatment groups differing only in ABT-450 dose (100 mg, 150 mg or 200 mg) were combined for safety analyses.
Measure: Number; unit: participants
Groups:
- Group A: Treatment-naïve participants received ABT-450 150 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 8 weeks.
- Group C + D: Treatment-naïve participants received ABT-450 (100 mg or 200 mg) and ritonavir 100 mg once daily, ABT-267 25 mg once daily, and ribavirin dosed by weight, twice daily, for 12 weeks.
- Group F + G: Treatment-naïve participants received ABT-450 (100 mg or 150 mg) and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 12 weeks.
- Group H + I: Treatment-naïve participants received ABT-450 (100 mg or 150 mg) and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 24 weeks.
- Group K + L: Participants who were null-responders to previous HCV treatment received ABT-450 (100 mg or 150 mg) and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 12 weeks.
- Group M + N: Participants who were null-responders to previous HCV treatment received ABT-450 (100 mg or 150 mg) and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 24 weeks.
Arm/Group | Group A | Group B | Group C + D | Group E | Group F + G | Group H + I | Group J | Group K + L | Group M + N
Number analyzed (Participants) | 80 | 41 | 79 | 79 | 79 | 80 | 45 | 45 | 45
participants
  Any adverse event | 67 | 36 | 71 | 68 | 71 | 77 | 42 | 39 | 37
  Any adverse event at least possibly DAA-related | 58 | 29 | 53 | 51 | 57 | 68 | 35 | 30 | 28
  Any severe adverse event | 3 | 0 | 3 | 5 | 3 | 3 | 1 | 1 | 1
  Any serious adverse event | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 0 | 2
  Any AE leading to discontinuation of study drug | 1 | 0 | 0 | 0 | 3 | 3 | 1 | 0 | 1
  Any AE leading to interruption of study drug | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0
  Any AE leading to ribavirin dose modification | 2 | 2 | 4 | 0 | 9 | 10 | 3 | 1 | 3
  Any fatal adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks Post-dose for 8 Weeks Versus 12 Weeks of Treatment With 3 DAAs and Ribavirin
Description: The percentage of participants achieving sustained virologic response 24 weeks after the last dose of study drug (SVR24), defined as hepatitis C virus (HCV) ribonucleic acid (RNA) less than the lower limit of quantitation (LLOQ), without any confirmed quantifiable (≥ LLOQ) post-treatment value before that time point. HCV RNA levels were measured from plasma by a central laboratory. The LLOQ for the assay was 25 IU/mL.
  The primary efficacy endpoint was the comparison between treatment-naïve participants following 8 weeks of treatment with 3 DAAs and ribavirin and those with 12 weeks of treatment with 3 DAAs and ribavirin (Group A versus Group G).
Time Frame: Post Treatment Week 24
Population: Intent-to-treat population (all participants who received at least 1 dose of direct-acting antiviral agent); participants with missing data were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Group A | Group B | Group C | Group D | Group E | Group F | Group G | Group H | Group I | Group J | Group K | Group L | Group M | Group N
Number analyzed (Participants) | 80 | 41 | 39 | 40 | 79 | 39 | 40 | 40 | 40 | 45 | 23 | 22 | 23 | 20
percentage of participants | 87.5 | 82.9 | 84.6 | 92.5 | 88.6 | 97.4 | 95.0 | 92.5 | 90.0 | 88.9 | 91.3 | 95.5 | 91.3 | 100.0
Statistical Analysis 1: Comparison: Group A vs Group G; The primary efficacy endpoint was the comparison of the percentage of treatment-naïve participants with SVR24 after treatment with 3 DAAs (at the 150 mg ABT-450 dose) and ribavirin for 8 weeks (Group A) versus 12 weeks (Group G). Logistic regression with baseline log10 HCV RNA level, treatment group, Interleukin 28B genotype (CC or non-CC), HCV subgenotype (1a or non-1a), and geographic region (US or non-US) as predictors; Test type: Superiority or Other; p = 0.406, Regression, Logistic — No adjustment for multiple comparison. Pre-specified 2-sided significance level of 0.05; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.09 to 2.61] — Odds ratio: Group A : Group G

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks Post-dose Following Treatment of Different Durations With 3 Direct-acting Antiviral Agents (DAAs) and Ribavirin
Description: This outcome measure compares the percentage of participants achieving sustained virologic response 24 weeks after the last dose of study drug (HCV RNA < LLOQ at post-treatment Week 24) following treatment with 3 DAAs (ABT-450/ritonavir, ABT-267, and ABT-333) and ribavirin in both treatment naïve and null-responder participants for 8 weeks (Group A) versus 12 weeks (Groups F + G + K + L) versus 24 weeks (Groups H + I + M + N).
Time Frame: Post-Treatment Week 24
Population: Intent-to-treat population; participants with missing data were counted as non-responders.
Measure: Number; unit: percentage of participants
Groups:
- Groups F + G + K + L: Participants (treatment-naïve and null-responders) received ABT-450 (100 mg or 150 mg) and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 12 weeks.
- Groups H + I + M + N: Participants (treatment-naïve and null-responders) received ABT-450 (100 mg or 150 mg) and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 24 weeks.
Arm/Group | Group A | Groups F + G + K + L | Groups H + I + M + N
Number analyzed (Participants) | 80 | 124 | 123
percentage of participants | 87.5 | 95.2 | 92.7
Statistical Analysis 1: Comparison: Group A vs Groups F + G + K + L; The percentage of participants with SVR24 after treatment for 8 weeks versus 12 weeks was compared using logistic regression with treatment group, baseline log10 HCV RNA level, HCV subgenotype (1a or non-1a), geographic region (US or non-US), Interleukin 28B genotype (CC or non-CC), and ABT-450/ritonavir dose and population (treatment-naïve or null-responders) as predictors; Test type: Superiority or Other; p = 0.266, Regression, Logistic — No adjustment for multiple comparison. Pre-specified 2-sided significance level of 0.05; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.08 to 2.02] — Odds ratio: Group A : Groups [F + G + K + L]
Statistical Analysis 2: Comparison: Group A vs Groups H + I + M + N; The percentage of participants with SVR24 after treatment for 8 weeks versus 24 weeks was compared using logistic regression with treatment group, baseline log10 HCV RNA level, HCV subgenotype (1a or non-1a), geographic region (US or non-US), Interleukin 28B genotype (CC or non-CC), ABT-450/ritonavir dose and population (treatment-naïve or null-responders) as predictors; Test type: Superiority or Other; p = 0.525, Regression, Logistic — No adjustment for multiple comparison. Pre-specified 2-sided significance level of 0.05; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.18 to 2.40] — Odds ratio: Group A : Groups [H + I + M + N]
Statistical Analysis 3: Comparison: Groups F + G + K + L vs Groups H + I + M + N; The percentage of participants with SVR24 after treatment for 12 weeks versus 24 weeks was compared using logistic regression with treatment group, baseline log10 HCV RNA level, HCV subgenotype (1a or non-1a), geographic region (US or non-US), Interleukin 28B genotype (CC or non-CC), ABT-450/ritonavir dose and population (treatment-naïve or null-responders) as predictors; Test type: Superiority or Other; p = 0.375, Regression, Logistic — No adjustment for multiple comparison. Pre-specified 2-sided significance level of 0.05; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.55 to 4.92] — Odds ratio: Groups [F + G + K + L] : Groups [H + I + M + N]

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks Post-dose Following Treatment for 12 Weeks With 2 DAAs and Ribavirin Versus 3 DAAs and Ribavirin
Description: This outcome measure compares the percentage of participants achieving sustained virologic response 24 weeks post-dose (HCV RNA < LLOQ at post-treatment Week 24) following treatment with 2 DAAs (ABT-450/ritonavir plus ABT-333 [Group B] or ABT-450/ritonavir plus ABT-267 [Groups C + D + J]) and ribavirin versus 3 DAAs (ABT-450/ritonavir plus ABT-333 and ABT-267) and ribavirin (Groups F + G + K + L).
Time Frame: Post-Treatment Week 24
Population: Intent-to-treat population; participants with missing data were counted as non-responders.
Measure: Number; unit: percentage of participants
Groups:
- Group B: Treatment-naïve participants received ABT-450 150 mg and ritonavir 100 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 12 weeks.
- Groups C + D + J: Participants (treatment-naïve and null-responders) received ABT-450 (100 mg or 200 mg) and ritonavir 100 mg once daily, ABT-267 25 mg once daily, and ribavirin dosed by weight, twice daily, for 12 weeks.
Arm/Group | Group B | Groups C + D + J | Groups F + G + K + L
Number analyzed (Participants) | 41 | 124 | 124
percentage of participants | 82.9 | 88.7 | 95.2
Statistical Analysis 1: Comparison: Group B vs Groups F + G + K + L; The percentage of participants with SVR24 after treatment with 2 DAAs and ribavirin versus 3 DAAs and ribavirin was compared using stratum-adjusted Mantel-Haenszel (MH) method with Interleukin 28B genotype (CC or non-CC) and HCV subgenotype (1a or non-1a); Test type: Superiority or Other; p = 0.068, Mantel Haenszel — No adjustment for multiple comparison. Pre-specified 2-sided significance level of 0.05; The Mantel-Haenszel method was used because logistic regression failed due to separation or quasi-separation; Difference = -12.16, 95% CI 2-sided [-25.20 to 0.88] — Difference = Group B - Groups [F + G + K + L]
Statistical Analysis 2: Comparison: Groups C + D + J vs Groups F + G + K + L; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.065, Mantel Haenszel — No adjustment for multiple comparison. Pre-specified 2-sided significance level of 0.05; The Mantel-Haenszel method was used because logistic regression failed due to separation or quasi-separation; Difference = -6.75, 95% CI 2-sided [-13.93 to 0.43] — Difference = Groups [C + D + J] - Groups [F + G + K + L]

5. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks Post-dose Following Treatment for 12 Weeks With 3 DAAs With Versus Without Ribavirin
Description: This outcome measure compares the percentage of participants achieving sustained virologic response 24 weeks post-dose (HCV RNA < LLOQ at post-treatment Week 24) following treatment with 3 DAAs with or without ribavirin (Group E versus Groups F + G + K + L).
Time Frame: Post-Treatment Week 24
Population: Intent-to-treat population; participants with missing data were counted as non-responders.
Measure: Number; unit: percentage of participants
Groups:
- Group E: Treatment-naïve participants received ABT-450 150 mg and ritonavir 100 mg once daily, ABT-267 25 mg once daily, and ABT-333 400 mg twice daily, for 12 weeks.
Arm/Group | Group E | Groups F + G + K + L
Number analyzed (Participants) | 79 | 124
percentage of participants | 88.6 | 95.2
Statistical Analysis 1: Comparison: Group E vs Groups F + G + K + L; The percentage of participants with SVR24 after treatment with 3 DAAs with and without ribavirin was compared using a stratum-adjusted Mantel-Haenszel (MH) method with Interleukin 28B genotype (CC or non-CC) and HCV subgenotype (1a or non-1a); Test type: Superiority or Other; p = 0.106, Mantel Haenszel — No adjustment for multiple comparison. Pre-specified 2-sided significance level of 0.05; The Mantel-Haenszel method was used because logistic regression failed due to separation or quasi-separation; Difference = -7.13, 95% CI 2-sided [-15.77 to 1.51] — Difference = Group E - Groups [F + G + K + L]

6. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks Post-dose in Treatment-naïve Versus Null-responders
Description: This outcome measure compares the percentage of participants achieving sustained virologic response 24 weeks post-dose (HCV RNA < LLOQ at post-treatment Week 24) following treatment with 3 DAAs and ribavirin in participants who were treatment-naïve versus those who were null-responders to previous HCV therapy (Groups F + G + H + I versus Groups K + L + M + N).
Time Frame: Post-Treatment Week 24
Population: Intent-to-treat population; participants with missing data were counted as non-responders.
Measure: Number; unit: percentage of participants
Groups:
- Groups F + G + H + I: Treatment-naïve participants received ABT-450 (100 mg or 150 mg) and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 12 or 24 weeks.
- Groups K + L + M + N: Participants who were null-responders to previous HCV treatment received ABT-450 (100 mg or 150 mg) and ritonavir 100 mg once daily, ABT-267 25 mg once daily, ABT-333 400 mg twice daily, and ribavirin dosed by weight, twice daily, for 12 or 24 weeks.
Arm/Group | Groups F + G + H + I | Groups K + L + M + N
Number analyzed (Participants) | 159 | 88
percentage of participants | 93.7 | 94.3
Statistical Analysis 1: Comparison: Groups F + G + H + I vs Groups K + L + M + N; The percentage of participants with SVR24 after treatment with 3 DAAs and ribavirin in treatment-naïve versus null-responders was compared using logistic regression with treatment group, baseline log10 HCV RNA level, HCV subgenotype (1a or non-1a), geographic region (US or non-US), Interleukin 28B genotype (CC or non-CC), and ABT-450/ritonavir dose as predictors; Test type: Superiority or Other; p = 0.616, Regression, Logistic — No adjustment for multiple comparison. Pre-specified 2-sided significance level of 0.05; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.37 to 5.34] — Odds ratio: Groups [F + G + H + I] : Groups [K + L + M + N]

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Description: Treatment groups differing only in ABT-450 dose (100 mg, 150 mg or 200 mg) were combined for safety analyses.
Arm/Group | Group A | Group B | Group C + D | Group E | Group F + G | Group H + I | Group J | Group K + L | Group M + N
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/41 | 2/79 | 2/79 | 1/79 | 1/80 | 0/45 | 0/45 | 2/43
Other Adverse Events (participants affected / at risk) | 64/80 | 33/41 | 66/79 | 59/79 | 66/79 | 74/80 | 40/45 | 36/45 | 34/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=80) | Group B (N=41) | Group C + D (N=79) | Group E (N=79) | Group F + G (N=79) | Group H + I (N=80) | Group J (N=45) | Group K + L (N=45) | Group M + N (N=43)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
FACIAL PARESIS (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
AFFECTIVE DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=80) | Group B (N=41) | Group C + D (N=79) | Group E (N=79) | Group F + G (N=79) | Group H + I (N=80) | Group J (N=45) | Group K + L (N=45) | Group M + N (N=43)
ANAEMIA (Blood and lymphatic system disorders) | 5 | 1 | 3 | 1 | 7 | 6 | 3 | 3 | 2
TINNITUS (Ear and labyrinth disorders) | 1 | 3 | 0 | 1 | 0 | 3 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 3 | 5 | 0 | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 3 | 4 | 3 | 3 | 7 | 1 | 6 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 2 | 5 | 3 | 4 | 4 | 0 | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 3 | 1 | 5 | 5 | 1 | 9 | 2 | 1 | 4
DIARRHOEA (Gastrointestinal disorders) | 8 | 10 | 8 | 13 | 10 | 11 | 7 | 8 | 8
DRY MOUTH (Gastrointestinal disorders) | 4 | 0 | 2 | 2 | 1 | 2 | 1 | 2 | 2
DYSPEPSIA (Gastrointestinal disorders) | 7 | 1 | 9 | 2 | 4 | 6 | 2 | 2 | 2
FLATULENCE (Gastrointestinal disorders) | 0 | 1 | 4 | 4 | 2 | 1 | 0 | 1 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 | 2 | 3 | 2 | 2 | 1 | 1 | 4
NAUSEA (Gastrointestinal disorders) | 12 | 7 | 16 | 11 | 19 | 20 | 6 | 9 | 8
VOMITING (Gastrointestinal disorders) | 7 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3
ASTHENIA (General disorders) | 7 | 1 | 8 | 5 | 3 | 12 | 10 | 4 | 4
CHEST PAIN (General disorders) | 0 | 1 | 2 | 0 | 1 | 4 | 1 | 3 | 0
CHILLS (General disorders) | 4 | 1 | 1 | 1 | 1 | 3 | 1 | 0 | 2
FATIGUE (General disorders) | 29 | 13 | 22 | 16 | 22 | 30 | 12 | 12 | 9
IRRITABILITY (General disorders) | 1 | 4 | 5 | 5 | 1 | 10 | 7 | 2 | 3
JAUNDICE (Hepatobiliary disorders) | 3 | 0 | 1 | 0 | 3 | 3 | 1 | 3 | 1
INFLUENZA (Infections and infestations) | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 3 | 0
NASOPHARYNGITIS (Infections and infestations) | 4 | 3 | 4 | 8 | 7 | 7 | 2 | 4 | 3
ORAL HERPES (Infections and infestations) | 2 | 0 | 2 | 2 | 1 | 3 | 3 | 3 | 2
RHINITIS (Infections and infestations) | 1 | 0 | 5 | 2 | 0 | 0 | 0 | 1 | 0
SINUSITIS (Infections and infestations) | 4 | 0 | 7 | 2 | 5 | 3 | 1 | 2 | 3
TOOTH INFECTION (Infections and infestations) | 2 | 0 | 0 | 1 | 4 | 4 | 1 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 1 | 5 | 5 | 4 | 5 | 3 | 4 | 0
URINARY TRACT INFECTION (Infections and infestations) | 4 | 3 | 2 | 1 | 0 | 6 | 2 | 3 | 2
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 8 | 1 | 5 | 3 | 3 | 6 | 3 | 1 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 2 | 6 | 7 | 5 | 8 | 3 | 5 | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 4 | 2 | 5 | 2 | 2 | 4
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 1 | 5 | 2 | 2 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 | 3 | 5 | 2 | 3 | 9 | 5 | 4 | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0 | 3 | 0 | 3 | 0
DISTURBANCE IN ATTENTION (Nervous system disorders) | 2 | 1 | 2 | 1 | 2 | 9 | 3 | 3 | 3
DIZZINESS (Nervous system disorders) | 5 | 7 | 2 | 4 | 3 | 8 | 4 | 1 | 4
DYSGEUSIA (Nervous system disorders) | 2 | 1 | 3 | 2 | 3 | 4 | 0 | 4 | 4
HEADACHE (Nervous system disorders) | 28 | 13 | 23 | 15 | 21 | 28 | 15 | 13 | 14
LETHARGY (Nervous system disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 3 | 2
MEMORY IMPAIRMENT (Nervous system disorders) | 0 | 0 | 1 | 3 | 0 | 5 | 1 | 0 | 2
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 3 | 1 | 1 | 2 | 1 | 0 | 5
ABNORMAL DREAMS (Psychiatric disorders) | 1 | 2 | 2 | 1 | 1 | 5 | 1 | 1 | 1
ANXIETY (Psychiatric disorders) | 2 | 2 | 0 | 3 | 4 | 6 | 4 | 1 | 3
DEPRESSED MOOD (Psychiatric disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 2 | 1
DEPRESSION (Psychiatric disorders) | 3 | 3 | 3 | 1 | 3 | 12 | 2 | 5 | 1
INSOMNIA (Psychiatric disorders) | 10 | 8 | 9 | 6 | 16 | 20 | 8 | 6 | 7
SLEEP DISORDER (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 11 | 2 | 8 | 12 | 7 | 3 | 9
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 4 | 1 | 5 | 8 | 4 | 3 | 3
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0 | 4 | 9 | 0 | 0 | 2
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4 | 0 | 1 | 4 | 2 | 4 | 2
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 6 | 0 | 0 | 4
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 | 3 | 3 | 1 | 4 | 6 | 6 | 4 | 4
PRURITUS (Skin and subcutaneous tissue disorders) | 12 | 3 | 8 | 3 | 6 | 11 | 6 | 7 | 6
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 2 | 5 | 0 | 1 | 4 | 3 | 5 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 10 | 2 | 6 | 6 | 11 | 15 | 2 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.